CLINICAL TRIAL: NCT06220162
Title: A Clinical Study of Chidamide in Combination With Venetoclax and Azacitidine (VAC) for Patients With Acute Myeloid Leukemia Who Did Not Achieve CR/CRi/MLFS (PR or NR) With One Cycle of Venetoclax and Azacitidine (VA).
Brief Title: VAC Regimen for AML Patients Who Failed to Response to VA Regimen
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Jining Medical University (Other); The Second People's Hospital of Huai'an (Other); The First Affiliated Hospital of Bengbu Medical University (Other); Northern Jiangsu People's Hospital (Other); Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, Prof., The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZAML04
Record Dates: First submitted 2024-01-06; First posted 2024-01-23 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML venetoclax azacitidine chidamide unfit
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; venetoclax; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VAC regimen (Experimental)
  Interventions: Drug: chidamide in combination with venetoclax and azacitidine (VAC)

INTERVENTIONS:
Drug: chidamide in combination with venetoclax and azacitidine (VAC) — Enrolled patients were given chidamide 10 mg every day on days 1-14, azacitidine 75mg/m2 every day on days 1-7, and oral venetoclax began at 100mg on day 1 and increased stepwise over 3 days to reach the target dose of 400mg (100mg, 200mg, and 400mg) on days 1-28. Dose adjustments for concomitant venetoclax with CYP3A4 inhibitors were made according to the literature.

SUMMARY:
Chidamide in combination with venetoclax and azacitidine (VAC) were expected to improve remission rate of patients following to VA regimen treatment failure.

DETAILED DESCRIPTION:
Venetoclax and azacitidine has become the standard first-line treatment for elderly/unsuitable AML patients who can't tolerate for intense chemotherapy.

However, a proportion of patients who were not able to achieve remission after failing to VA regimen and then were given the second cycle, and their rate of achieving remission was even lower. Chidamide down-regulates the expression of MCL and is expected to improve the remission rate further in combination with VA regimen.

ELIGIBILITY:
Inclusion Criteria:

Patients with AML who are not suitable for intensive chemotherapy according to the WHO diagnosis: age ≥60 years or age <60 years but fulfil the following criteria;

1. Age 18 to 59 years;
2. Eastern Cooperative Oncology Group (ECOG) physical status score of 2 or 3;
3. Expected survival time ≥3 months;
4. Or fulfilment of severe cardiac, pulmonary, hepatic, or renal disease; (A) Presence of a cardiac history of congestive heart failure, or ejection fraction ≤ 50%, or presence of chronic stable angina; (B) Lung carbon monoxide diffusing capacity (DLCO) ≤ 65%, or first forced expiratory volume (FEV1) ≤ 65%; (C) Moderate hepatic impairment with total bilirubin > 1.5 to ≤ 3.0 x upper limit of normal (ULN); (D) Creatinine clearance ≥ 30 mL/min to < 45 mL/min;
5. Not received radiotherapy, treatment regimens other than the VA regimen, or haematopoietic stem cell transplantation within 4 weeks prior to enrolment;
6. Other comorbidities that, in the judgement of the physician, make the administration of intensive chemotherapy unsuitable;
7. Ability to understand and willingness to sign the informed consent for this trial;
8. The patient refuses intensive chemotherapy and has the willingness to accept non-intensive chemotherapy.

Exclusion Criteria:

1. Patients with a history of myeloproliferative neoplasms (MPN), including myelofibrosis, thrombocythemia, polycythaemia vera, chronic granulocytic leukemia (CML) with or without BCR-ABL1 translocation, and AML or acute promyelocytic leukemia (APL) with BCR-ABL1 translocation;
2. Patients with FLT3 mutations and who were treated with targeted agents (inclusion is possible if the use of specific targeted agents is discontinued);
3. Patients with less than 50% reduction of blasts after VA regimen;
4. Patients with active CNS involvement;
5. With prior treatment with chidamide;
6. Clinically uncontrolled active infections (including bacterial, fungal or viral infections) and organ hemorrhage;
7. Pregnant or lactating women;
8. Participation in any other clinical trial within 3 months prior to VAC regimen;
9. With other malignant tumours;
10. With uncontrolled mental disorders;
11. Any other condition that, in the opinion of the investigator, makes it inappropriate to participate in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
ORR(overall response rate) | 1 month
  ORR was calculated as the sum of CR, CRi, MLFS and PR.

SECONDARY OUTCOMES:
OS (Overall survival) | 2 years
  OS was defined as the time from enrollment to this study to the date of death from any cause; patients not known to have died at last follow-up are censored on the date they were last known to be alive.
EFS (Event-free survival) | 2 years
  EFS was defined as the time from the initiation of CAV to treatment failure, relapse, death from any cause or the last follow-up.
Adverse events (AEs) | 2 months
  It is evaluated and graded according to CTCAE 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Li Xue, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No